CLINICAL TRIAL: NCT06889493
Title: A Phase 1 Trial of the Oncolytic Virus SVV-001 in Combination With Nivolumab and Ipilimumab in Patients With Poorly Differentiated Neuroendocrine Carcinomas or Well-Differentiated High-Grade (Grade 3) Neuroendocrine Tumors
Brief Title: SVV-001 With Nivolumab and Ipilimumab in Patients With Poorly Differentiated Neuroendocrine Carcinomas (NEC) or Well-Differentiated High-Grade Neuroendocrine Tumors (NET)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Peter Hosein, MD (Other)
Collaborators: Seneca Therapeutics (Unknown)
Responsible Party: Sponsor-Investigator, Peter Hosein, MD, Associate Professor of Clinical, University of Miami Sylvester Comprehensive Cancer Center
Organization: University of Miami (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20231325
Record Dates: First submitted 2025-03-15; First posted 2025-03-21 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Neuroendocrine Carcinoma; Neuroendocrine Tumors
MeSH Terms: conditions — Carcinoma, Neuroendocrine; Neuroendocrine Tumors | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SVV-001 Single Dose Treatment Group (Experimental): Participants in this group will receive a single dose of SVV-001 on Day 1, in combination with Nivolumab and Ipilimumab therapy.
  Total participation duration is up to 2 years.
  Interventions: Biological: Seneca Valley Virus-001 (SVV-001); Drug: Nivolumab; Drug: Ipilimumab
- SVV-001 Multi-Dose Treatment Group (Experimental): Participants in this group will receive multiple doses of SVV-001, beginning on Day 1, in combination with Nivolumab and Ipilimumab therapy.
  Total participation duration is up to 2 years.
  Interventions: Biological: Seneca Valley Virus-001 (SVV-001); Drug: Nivolumab; Drug: Ipilimumab
- SVV-001 RP2D Treatment Group (Experimental): Participants is this group will receive the recommended phase 2 dose and frequency of SVV-001 in combination with Nivolumab and Ipilimumab therapy.
  Total participation duration is up to 2 years.
  Interventions: Biological: Seneca Valley Virus-001 (SVV-001); Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Biological: Seneca Valley Virus-001 (SVV-001) — SVV-001 will be administered intratumorally as a single dose on Day 1; or as multiple doses on Days 1, 15, 29, 43, 57, and 71. The virus dose levels per SVV-001 treatment are as follows:
  * 2.2 × 10^8 Viral Genomes (VG) (starting dose)
  * 2.2 × 10^9 VG
  * 2.2 × 10^10 VG
Drug: Nivolumab — Nivolumab will be administered via intravenous (IV) injection at a dose of 240 mg, once every two weeks starting on Day 15 until Day 85 during SVV-001 therapy. Nivolumab will be administered once every four weeks during the maintenance period for up to 2 years.
Drug: Ipilimumab — Ipilimumab will be administered via intravenous (IV) injection at a dose of 1 mg/kg, once every six weeks starting on Day 15 until Day 85 during SVV-001 therapy. Participants will continue on 1 mg/kg ipilimumab IV every 6 weeks for two additional doses or unacceptable toxicity and/or participant withdrawal.

SUMMARY:
The purpose of this study is to determine:

1. The highest dose of the trial intervention that targets neuroendocrine tumors and is tolerated by patients.
2. The highest frequency of dosing of the trial intervention that targets neuroendocrine tumors and is tolerated by patients.
3. The highest dose and frequency of dosing of the trial intervention that targets neuroendocrine tumors with at least the same degree of effectiveness and tolerability as currently available (standard of care) treatments for patients with neuroendocrine tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, 18 years of age or older at the time of consent.
2. Life expectancy of 6 months or greater as assessed by the treating oncologist.
3. Have advanced metastatic disease that has progressed on at least one line of available therapy.
4. Histologically or cytologically confirmed diagnosis of Grade 3 well-differentiated neuroendocrine tumor (NET) or poorly differentiated neuroendocrine carcinoma (NEC; large-cell neuroendocrine carcinoma, small-cell carcinoma, mixed neuroendocrine non neuroendocrine carcinoma). Note: if an archival tissue sample collected ≤ 2 years from enrollment is unavailable at Screening for diagnostic confirmation, at the Principal Investigator's (PI's) discretion, a screening biopsy will be ordered.
5. For patients in Part 1A, in addition to histological or cytological confirmation of NEC or NET (see Inclusion #4), radiological confirmation of tumor is required.
6. Parts 1B and 2 only: Measurable disease as determined by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 or immune-related Response Evaluation Criteria in Solid Tumors (iRECIST). At least one lesion must be suitable for multiple injections (up to 6 injections every 2 weeks) with SVV-001. Lesions for injection must be ≥10 mm in longest diameter and deemed safe and suitable for injection by the Investigator.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
8. Recovered to Grade 1 or baseline from any clinically significant toxicity associated with prior treatments (excluding alopecia) prior to initiation of investigational medicinal product (IMP) administration.
9. Adequate hematological, renal, and liver function defined as follows:

   * a. Hepatic:

     * i. Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 × upper limit of normal (ULN) (≤5 × ULN if liver metastases are present)
     * ii. Serum bilirubin ≤1.5 × ULN (unless due to Gilbert's syndrome or hemolysis)
   * b. Renal:

     * i. Creatinine clearance ≥50 mL/minute using Cockcroft Gault equation
   * c. Hematologic:

     * i. Absolute neutrophil count ≥1500 cells/µL
     * ii. Platelet count ≥100,000 platelets/µL
     * iii. Hemoglobin ≥9.0 g/dL
     * iv. International normalization ratio (INR) within the institutional normal range
     * v. Normal prothrombin time (PT) and partial thromboplastin time (PTT)
10. For Part 2 Expansion Cohort patients only, patients will submit archival tissue at Screening and undergo a post-treatment biopsy according to the treating institution's guidelines with the following exceptions:

    * a. If an archival tissue sample collected ≤ 2 years from enrollment is unavailable at Screening, at the PI's discretion, a screening biopsy will be ordered.
    * b. Participants will not undergo a biopsy procedure for collection of the post-treatment biopsy if, in the discretion of their treating physician, the participant's condition has deteriorated to the point where performance of a biopsy procedure would place the participant at an increased risk for complications beyond what is reasonably expected for a biopsy collected as part of the participant's standard medical care.
11. Women of childbearing potential must agree to use a reliable form of contraceptive during the trial treatment period and for at least 7 months following the last dose of IMP.
12. Male patients must agree to use an adequate method of contraception during the trial treatment period and for at least 7 months following the last dose of IMP.
13. Patient is willing and able to comply with all protocol-required assessments, visits, and procedures.
14. Provide written informed consent prior to performing any trial-related procedure.

Exclusion Criteria:

1. Any active second malignancy within the 2 years prior to the screening visit, unless the patient has undergone curative surgery for the tumors such as in situ cervical cancer or squamous cell cancer of the skin.
2. Has had cytotoxic chemotherapy or radiation therapy within 3 weeks; and less than 5 half-lives or 6 weeks, whichever is shorter, from prior biologic therapies, prior to the first dose of SVV-001.
3. Has undergone a major surgical procedure (as defined by the Investigator) or significant traumatic injury within 28 days prior to the first dose of SVV-001.
4. Has any physical abnormality of the tissue/organ to be biopsied that would put the patient at increased risk of bleeding secondary to the injection and/or biopsy.
5. Has received a live-virus immunization within 30 days prior to the screening visit or anticipates receiving a live virus immunization during the trial or within 30 days of the last treatment with IMP.
6. Presence of an active autoimmune or inflammatory disease requiring systemic treatment within the past 2 months or a documented history of clinically severe autoimmune disease that requires systemic steroids or other immunosuppressive medications. Local steroid injections, intermittent use of topical, inhaled, ophthalmologic, intra-articular, or intranasal corticosteroids, or systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or equivalent would not result in exclusion from the trial.
7. Presence of primary immunodeficiency or receiving systemic steroids of >10 mg/day prednisone or equivalent or other immunosuppressive agents within 14 days prior to the first dose of SVV-001.
8. Any active infection, including known infection with human immunodeficiency virus (HIV), active hepatitis, or seropositive for hepatis B immunoglobulin (Ig) M core antibody or hepatitis C ribonucleic acid (RNA) at the screening visit.
9. Patients with a history of solid-organ or bone marrow transplant.
10. Known hypersensitivity to ipilimumab or nivolumab or their excipients
11. Has known untreated central nervous system metastases. Patients with treated brain metastases are eligible as long as they are stable and there is no evidence of progression for at least 4 weeks after central nervous system-directed treatment, as ascertained by clinical examination and brain imaging (magnetic resonance imaging (MRI) or computed tomography (CT)) during the screening period.
12. Any clinically significant (i.e., active) cardiovascular disease, including cerebral vascular accident/stroke (<6 months prior to enrollment), myocardial infarction (<6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication.
13. Patients with an ejection fraction (EF) < 50 on a 2D echocardiogram (ECHO).
14. Patients whose baseline pulse oximetry (saturation of peripheral oxygen (SpO2)) is < 92% on Room air.
15. Any chronic illness, psychiatric condition, or social situation that is life threatening or, in the opinion of the Investigator, renders the patient unsuitable for participation in a clinical trial due to possible noncompliance or would place the patient at an unacceptable risk and/or have the potential to affect interpretation of the results of the trial.
16. Female participants who are breastfeeding and/or who have a positive pregnancy test result prior to receiving any treatment with IMP.
17. Patients with impaired decision-making capacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2030-06-01 (Estimated); Study Completion 2030-06-01 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD)/Recommended Phase 2 Dose | Up to 12 months
  MTD is defined as the highest dose of SVV-001 evaluated for which estimated toxicity rate is the closest to the target toxicity rate as assessed by treating physician using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. The MTD will be established as the recommended phase 2 dose (RP2D).
Number of Participants Experiencing Dose Limiting Toxicities (DLTs): Part 1 Only | Up to 12 months
  The number of participants experiencing dose limiting toxicities (DLTs) in Part 1 will be reported. DLTs will be assessed using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, per physician discretion.
Number of Participants Experiencing Treatment-Related Serious Adverse Events (SAEs) | Up to 12 months
  The number of participants experiencing treatment-related serious adverse events (SAEs) after starting study therapy will be reported. SAEs will be assessed using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, per physician discretion.
Number of Participants Experiencing Treatment-Related Adverse Events (AEs) | Up to 12 months
  The number of participants experiencing treatment-related adverse events after starting study therapy will be reported. AEs will be assessed using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, per physician discretion.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) Measured by RECIST | Up to 12 months
  Progression-Free Survival (PFS) among study participants will be reported. PFS will be assessed in months (6 and 12 months) from start of treatment according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
Progression-Free Survival (PFS) Measured by iRECIST | Up to 12 months
  Progression-Free Survival (PFS) among study participants will be reported. PFS will be assessed in months (6 and 12 months) from start of treatment according to immune-related Response Evaluation Criteria in Solid Tumors (iRECIST).
Overall Response Rate (ORR) Measured by RECIST | Up to 12 months
  ORR is defined as percentage of evaluable patients achieving complete response (CR) or partial response (PR), as best responses according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
Overall Response Rate (ORR) Measured by iRECIST | Up to 12 months
  ORR is defined as percentage of evaluable patients achieving complete response (CR) or partial response (PR), as best responses according to immune-related Response Evaluation Criteria in Solid Tumors (iRECIST).
Duration of Response (DOR) | Up to 2 years
  Duration of overall response is defined as time in months from date of onset of response (the first documentation of partial response (PR) or complete response (CR)) to the date of first disease progression after initiation to study therapy.
Clinical Benefit Rate (CBR) Measured by RECIST | Up to 12 months
  Clinical benefit rate (CBR) is defined as percentage of evaluable patients achieving complete response (CR) or partial response (PR) or stable disease (SD) as best response, according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
Clinical Benefit Rate (CBR) Measured by iRECIST | Up to 12 months
  Clinical benefit rate (CBR) is defined as percentage of evaluable patients achieving complete response (CR) or partial response (PR) or stable disease (SD) as best response, according to immune-related Response Evaluation Criteria in Solid Tumors (iRECIST).

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hosein, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No